CLINICAL TRIAL: NCT04927390
Title: A Randomised Prospective Open Label Pilot Trial Comparing Mycophenolate Mofetil (MMF) With no Immunosuppression in Adults With Limited Cutaneous Systemic Sclerosis
Brief Title: Mycophenolate in Limited Cutaneous Systemic Sclerosis (MINIMISE-Pilot)
Acronym: MINIMISE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University College, London (Other)
Collaborators: Versus Arthritis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTU/2017/306; 2019-004139-21 (EudraCT Number)
Record Dates: First submitted 2021-05-19; First posted 2021-06-16 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Systemic Sclerosis; Limited Cutaneous Systemic Sclerosis
Keywords: Limited Cutaneous Systemic Sclerosis; Mycophenolate Mofetil
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Limited | interventions — Mycophenolic Acid

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomised 1:1 to receive Mycophenolate Mofetil plus Standard of Care (MMF Group) or Standard of Care alone (Control Group).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mycophenolate Mofetil (MMF) Arm (Experimental): Participants will receive mycophenolate mofetil (MMF) for up to 96 weeks, in addition to their background Standard of Care medication for systemic sclerosis related symptoms. They will receive 500mg twice daily over the first 4 weeks following their randomisation, and if tolerated the dose will be increased to a target dose of 1g twice daily starting from week 5 until their Final visit.
  Interventions: Drug: Mycophenolate Mofetil 500mg
- Control Arm (No Intervention): Standard of Care (no immunosuppression) for systemic sclerosis related symptoms.

INTERVENTIONS:
Drug: Mycophenolate Mofetil 500mg — Mycophenolate Mofetil oral tablet twice daily for up to 96 weeks
  Arms: Mycophenolate Mofetil (MMF) Arm

SUMMARY:
Systemic sclerosis or scleroderma is an autoimmune condition that cause thickening and hardening of the skin, but can also affect internal organs. There are two major subsets of scleroderma: the limited cutaneous systemic sclerosis (lcSSc) that usually affects the skin of the face, neck, lower legs or lower arms, but can also lead to internal organ complications, and the diffuse cutaneous systemic sclerosis (dcSSc) that may affect blood circulation and internal organs, as well as the skin. To date there is no drug that has been definitively proven to cure or modify the course of scleroderma. However, there is emerging evidence that immunosuppression and specifically mycophenolate mofetil (MMF) may be beneficial in lcSSc.

The MINIMISE-Pilot trial would be an important first step to evaluate the risk and potential benefit to this disease group. MMF as the intervention of choice is both appropriate and timely, as it has been routinely used in the management of dcSSc. The aim of this pilot trial is to explore whether the immunosuppressive agent MMF can slow down disease progression in patients with lcSSc compared to the current standard of care alone. This pilot trial will also provide critical information for the development of a future large trial that could potentially transform lcSSc patient management.

DETAILED DESCRIPTION:
The MINIMISE-Pilot trial aims to explore whether the immunosuppressive agent mycophenolate mofetil (MMF) at a target dose of 2g daily can slow down disease progression in patients with limited cutaneous systemic sclerosis (lcSSc) compared to the current standard of care alone. This pilot trial will also provide critical information for the development of a future large trial that could potentially transform lcSSc patient management.

This is an open label randomised prospective trial that will recruit 120 participants aged 18 and older with limited cutaneous systemic sclerosis across 13 sites in the UK. Following a screening visit, eligible participants will attend a baseline visit where they will be randomly allocated into one of two groups; MMF or Control. Those in the first group are given mycophenolate mofetil (MMF) taken daily by mouth for up to 96 weeks, in addition to their background Standard of Care medication for SSc related symptoms. Those in the second group will not receive any MMF but will remain on their standard of care medication alone.

Participants are expected to be followed up for a minimum of 48 weeks or a maximum of 96 weeks. The trial will involve five (5) clinic visits which are expected to be carried out at the same time of the participants' normal hospital appointment with their scleroderma specialist. Participants from both groups will have the same assessments. Participants are expected to return to the clinics at Week 24, 48, 72 and 96. However, participants allocated to the MMF group will have additional blood samples taken for safety monitoring every 2 weeks for the first 8 weeks, then every 4 weeks for the following 12 weeks. Thereafter, every 12 weeks up to their final visit.

All the participants will receive four (4) routine telephone calls in between their clinic visits.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with lcSSc classified by the 2013 EULAR ACR criteria for limited cutaneous subset of SSc
2. Participants with less than 7 years disease duration from first non-Raynaud's manifestation of SSc
3. Participants aged 18 years or more (≥ 18 years) at screening visit
4. If women of child bearing potential, the participant must have a negative pregnancy test at screening and baseline visits
5. Negative viral screen for HIV, Hepatitis B and C
6. Ability to provide full informed consent
7. Registered with a GP practice in the UK
8. Participants must be willing to attend for follow up visits (at site or remotely) and to comply with study-related procedures -

Exclusion Criteria:

1. Having already developed a complication of SSc that requires initiation of MMF or an alternative major immunosuppressive drug for SSc such as methotrexate, cyclophosphamide or azathioprine
2. Treatment with methotrexate, cyclosporine A, azathioprine, mycophenolate mofetil (MMF), rapamycin, colchicine, D-penicillamine, within ≤ 4 weeks prior to the baseline visit date
3. Contraindication to MMF (e.g. active infection that would preclude MMF in judgement of investigator), or previous intolerance of MMF
4. Any clinical condition which the investigator considers would make the patient unsuitable for the trial
5. Pregnancy (or planned pregnancy during trial participation) and/or breastfeeding
6. Women of child bearing potential and male participants with a partner of child bearing potential not willing to use adequate contraception as described in section 6.3.1.4 for the duration of trial treatment and within the time points specified following last trial treatment.
7. Active chronic infection such as COVID-19, tuberculosis, pneumocystis, cytomegalovirus, herpes simplex virus, herpes zoster and atypical mycobacteria.

   Suitability for enrolment once the participant has recovered from infection will be based on Investigator judgment.
8. Infection history:

   i. Hospitalisation for treatment of infection within ≤ 8 weeks of screening visit date

   ii. Use of parenteral (IV or IM) antibiotics (antibacterials, antivirals, anti-fungals, or anti-parasitic agents) within ≤ 4 weeks of screening visit date
9. Receipt of a live-attenuated vaccine within ≤ 12 weeks of screening visit date
10. Participants enrolled in any other interventional trial within ≤ 4 weeks of the screening visit date (co-enrolment in observational studies is acceptable)
11. Current drug or alcohol abuse or dependence, or a history of drug or alcohol abuse or dependence within ≤ 52 weeks prior to screening visit date.
12. Any of the following laboratory results at screening visit:

    * Glomerular filtration rate (GFR) <60 ml/min/1.73m²
    * Absolute neutrophil count (ANC) < 1.6 x 10^9/l
    * ALT or AST > 2 x ULN
13. Participants not willing or unable to attend on-site screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-12-08 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
The total number of lcSSc patients screened during the 12 month recruitment period, measured from information provided on the site Screening Logs | From first site activation up to a period of 12 months
  The total number of lcSSc patients screened will be captured on detailed screening logs
The proportion of participants who provide consent during the 12 month recruitment period, measured from information provided on the site Screening Logs | From first site activation up to a period of 12 months
  Participant informed consent will be captured in detailed screening logs
The proportion of participants who meet the eligibility criteria during the 12 month recruitment period, measured from information provided on the site Screening Logs | From first site activation up to a period of 12 months
  Information on participants who meet the eligibility criteria will be captured on detailed screening logs
Adherence to trial treatment by participants randomised to the MMF arm as assessed by the Participant Dosing Diaries. | From Baseline, up until a minimum of 48 weeks or a maximum of 96 weeks
  Participant self-reported adherence using participant dosing diaries to be completed daily. Diaries will be provided to all participants randomised to MMF to record their daily trial medication intake, in addition to any dose modifications and dose interruptions for the duration of their time in the study.
Drug adherence rate from participants randomised to the MMF arm, measured by Pharmacy Accountability Logs | From first participant dispensing, through study completion up to 36 months
  Pharmacy dispensing accountability logs will record the number of pills dispensed at each visit and the number of pills returned by the participant.(i.e. pill count)
  The number of pills taken is calculated by subtracting the count of the number of pills remaining from the total number of pills dispensed. The drug adherence rate is then calculated by dividing the number of pills taken by number of days elapsed since the last dispense.
Adherence to the study protocol by participating sites as assessed by the number of protocol deviations reported using the Protocol Deviation Reports | From Screening, through study completion up to 36 months
  Sites to report deviations and sponsor protocol compliance reviews during central, remote and on-site monitoring to be reported in Protocol Deviation Reports.
The proportion of participants intolerant to MMF who discontinue trial treatment from Baseline for a minimum of 48 weeks or a maximum of 96 weeks as assessed by the Participant withdrawal Logs | From Baseline, up until a minimum of 48 weeks or a maximum of 96 weeks
  The number of participants who withdraw from trial treatment ONLY will be recorded using detailed Participant Withdrawal Logs
The total number of participants randomised to MMF who reach the target dose of 2g a day, measured by medication intake information captured in the Participant Dosing Diaries | From Baseline through to study completion for a minimum of 48 weeks or a maximum of 96 weeks
  Self-reported: Participant Dosing Diaries will be provided to all participants randomised to MMF to record dose escalation information and daily intake of the IMP .
The total number of participants randomised to MMF and Control who reach a clinical worsening of disease progression, measured by the modified Rodnan Skin Score (mRSS) from Baseline, every 6 months until Final trial visit. | From Baseline, every 6 months, through study completion up until a minimum of 48 weeks or a maximum of 96 weeks
  Validated physical examination method for estimating skin induration. It is scored on a 0 (normal) to 3+ (severe induration) ordinal scales over 17 body areas, with a maximum score of 51 and is used to categorise severity of SSc. Minimally clinically significant difference in mRSS is 3-5 points.
  The measurement of time to clinically important disease progression will demonstrate a clinically important advantage of active treatment compared with no immunosuppression if a beneficial effect is found.
The number of participant loss to follow- up as assessed by the Participant Withdrawal Logs | From Baseline, through study completion up until a minimum of 48 weeks or a maximum of 96 weeks
  The number of participant loss to follow -up in each group (MMF or control) will be recorded using detailed Participant Withdrawal Logs

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 from Baseline for a minimum of 48 weeks or a maximum of 96 weeks | From Baseline, through study completion for a minimum of 48 weeks or a maximum of 96 weeks
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 from Baseline for a minimum of 48 weeks or a maximum of 96 weeks
Number of reported deaths Baseline | From Baseline , through study completion, up to 36 months
  Participants self report, review of hospital records
Changes in functional ability from Baseline for a minimum of 48 weeks or a maximum of 96 weeks as measured by the Scleroderma Assessment Questionnaire | From Baseline, every 6 months, through study completion up until a minimum of 48 weeks or a maximum of 96 weeks
  The Scleroderma Assessment Questionnaire is a self-assessed measure ranging from 0-3 (where 0 = without difficulty and 3 = unable to do) for several questions including vascular, respiratory, gastrointestinal, musculoskeletal, and overall disease status with 23 questions divided into 4 groups.
Quality of Life as measured by the EQ5-5D-5L Questionnaire from Baseline for a minimum of 48 weeks or a maximum of 96 weeks | From Baseline, every 6 months, through study completion up until a minimum of 48 weeks or a maximum of 96 weeks
  EQ-5D- 5L is a participant self -reported questionnaire which evaluates the generic quality of life at the time of completion. It comprises of one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
  Respondents are asked to choose the statement in each dimension that best describes their health status. Their responses are coded as a number (1, 2, or 3) that corresponds to the respective level of severity: 1 indicates no problems, 2 some problems, and 3 extreme problems
Changes in pain and disability from Baseline for a minimum of 48 weeks or a maximum of 96 weeks as measured by the Patient Global Questionnaire. | From Baseline, every 6 months, through study completion up until a minimum of 48 weeks or a maximum of 96 weeks
  Self-reported questionnaire assessed by a single question to reflect the participants perspective on their health overall. Rating scale used with a 0-100 response, where 0= has no effect at all, 100= worst possible effect.
Changes in pain and disability from Baseline for a minimum of 48 weeks or a maximum of 96 weeks as measured by the Physician's Global Questionnaire. | From Baseline, every 6 months, through study completion up until a minimum of 48 weeks or a maximum of 96 weeks]
  Physician-reported questionnaire assessed by a single question to reflect the participants perspective on their health overall. Rating scale used with a 0-100 response, where 0= has no effect at all, 100= worst possible effect.
Scleroderma skin activity and skin-related health related quality of life from Baseline for a minimum of 48 weeks or a maximum of 96 weeks as measured by PASTUL-SSPRO score | From Baseline, every 6 months, through study completion up until a minimum of 48 weeks or a maximum of 96 weeks
  Self-reported questionnaire specifies a grading of skin (normal (0), mild (1), moderate (2), severely (3) thickened) at eight sites corresponding to mRSS with maximum score assigned to each site (PASTUL), and that assesses health-related quality of life (HRQOL) related to skin involvement in SSc. It has 18 items representing 4 HRQOL scales: physical effects, emotional effects, physical function, and social effects. All items are scored from 0 (better) to 6 (worse) (SSPRO).

OTHER OUTCOMES:
Subgroup analyses of antinuclear antibody, ACA+ versus ACA- | over 36 months
  Standard diagnostic laboratory assays for antinuclear antibodies
IcSSc disease duration at baseline | Baseline
  IcSSc disease duration at baseline up to 4 years versus four years or more

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Denton, Principal Investigator — University College, London
Locations (12):
- United Kingdom (12):
  - Royal United Hospitals Bath Nhs Foundation Trust, Bath
  - Southmead Hospital - NORTH BRISTOL NHS TRUST, Bristol
  - Darlington Memorial Hospital - County Durham and Darlington NHS Foundation Trust, Darlington
  - Ninewells Hospital - NHS Tayside, Dundee
  - Chapel Allerton Hospital - LEEDS TEACHING HOSPITALS NHS TRUST, Leeds
  - Aintree University Hospital NHS Foundation Trust, Liverpool
  - Royal Free Hospital - Royal Free NHS Foundation Trust, London
  - Manchester Royal Infirmary - Manchester University NHS Foundation Trust, Manchester
  - Salford Hospital - Northern Care Alliance NHS Foundation Trust, Manchester
  - Freeman Hospital - THE NEWCASTLE UPON TYNE HOSPITALS NHS FOUNDATION TRUST, Newcastle
  - Royal Hallamshire Hospital - SHEFFIELD TEACHING HOSPITALS NHS FOUNDATION TRUST, Sheffield
  - The Royal Wolverhampton Nhs Trust, Wolverhampton

IPD SHARING:
Plan to Share IPD: Undecided
No plan to share IPD has been made at this time

REFERENCES:
- See also: Sponsor website link to trial — https://www.ucl.ac.uk/comprehensive-clinical-trials-unit/research-projects/2020/may/minimise